CLINICAL TRIAL: NCT00401713
Title: Transplantation of Autologous RPE Versus Translocation of Autologous RPE and Choroid in AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Univ Prof Dr Susanne Binder, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR-01-CI-2006
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: submacular membrane; transplantation of RPE; translocation of RPE and Choroid
MeSH Terms: conditions — Macular Degeneration

INTERVENTIONS:
Procedure: Transplantation of autologous RPE — RPE cell suspension
Procedure: Translocation of autologous RPE and Choroid — RPE patch

SUMMARY:
The purpose of this study is to evaluate two surgical interventions in patients with AMD.

DETAILED DESCRIPTION:
The Submacular surgical trials have shown that submacular membrane extraction alone did not improve or preserve visual acuity in patients with AMD. Transplantation of autologous RPE and translocation of autologous RPE and choroid represent two promising therapeutic interventions in patients with AMD. This prospective, randomized clinical trial compares the two surgical treatments and additionally compares the clinical results (visual acuity, FLA) with OCT- and UHR-OCT data.

ELIGIBILITY:
Inclusion Criteria:

* AMD and submacular cnv
* non responders to laser treatment or pdt
* treatment: rpe transplantation or rpe + choroid translocation
* age over 50 years

Exclusion Criteria:

* other additional retinal diseases, like diabetic or hypertensive retinopathy and vascular diseases.
* optic atrophy
* unstable glaucoma

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Visual Acuity: distance and near | preoperatively, 1 months, 3 months, 12 months, +/- 18 months, 36 months
FLA | (preoperatively, 3 months, +/- 12 months after surgery)

SECONDARY OUTCOMES:
OCT | (preoperatively, 3 months, 12 months after surgery)
UHR OCT | (after surgery, including silicone oil removal)
autofluorescence | (preoperatively, 3 months, +/- 12 months after surgery)
perimetry | (if feasible)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, MD, Principal Investigator — Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery, Department of Ophthalmology, Rudolf Foundation Clinic
Locations (1):
- Department of Opthalmology, Rudolf Foundation Clinic, Vienna, Vienna, Austria

REFERENCES:
- [Background] van Meurs JC et al Br J opthalmol 2004; 88:110-113
- [Background] van Meurs JC, Van Den Biesen PR. Autologous retinal pigment epithelium and choroid translocation in patients with exudative age-related macular degeneration: short-term follow-up. Am J Ophthalmol. 2003 Oct;136(4):688-95. doi: 10.1016/s0002-9394(03)00384-2. PMID 14516809
- [Derived] Falkner-Radler CI, Krebs I, Glittenberg C, Povazay B, Drexler W, Graf A, Binder S. Human retinal pigment epithelium (RPE) transplantation: outcome after autologous RPE-choroid sheet and RPE cell-suspension in a randomised clinical study. Br J Ophthalmol. 2011 Mar;95(3):370-5. doi: 10.1136/bjo.2009.176305. Epub 2010 Jul 7. PMID 20610478